CLINICAL TRIAL: NCT00001983
Title: Screening Protocol to Evaluate Patients for Approved Studies
Brief Title: Eligibility Screening for National Institute of Dental and Craniofacial Research Studies
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000066; 00-D-0066
Record Dates: First submitted 2000-01-26; First posted 2000-01-27 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-12

CONDITIONS: Fibromyalgia
Keywords: Questionnaires; Eligibility; History; Physical Examination; Tests; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

SUMMARY:
This screening protocol is designed to evaluate patients for participation in clinical studies in the Gene Therapy and Therapeutics Branch (GTTB) of the National Institute of Dental and Craniofacial Research. To participate, patients must meet the specific requirements of at least one of the available research studies; this protocol serves as a first step for admitting patients to an appropriate program.

People with diagnosed or undiagnosed conditions may participate in this screening protocol. They will undergo procedures that may include questionnaires, a physical examination, routine laboratory tests, and diagnostic imaging or radiological studies. Eligibility screening will be limited to three visits within 12 months of entry into the protocol. If an appropriate study is not found by the end of this time, the candidate's participation in the screening program will terminate. No experimental treatments are offered under the screening protocol.

Patients who are found eligible for a current GTTB study will be notified of their options and invited to enroll.

DETAILED DESCRIPTION:
This protocol is designed to screen patients with either diagnosed or undiagnosed conditions, and provides for determining eligibility for approved protocols within the Gene Therapy and Therapeutics Branch (GTTB), National Institute of Dental and Craniofacial Research. The purpose of the protocol is to allow evaluation of patients who do not meet the requirements for other screening protocols, such as the screening protocol for Sjogren's syndrome patients.

Each subject will be evaluated to determine whether they are suitable candidates for inclusion in any protocols in the GTTB. The screening evaluation will include past and current medical history, and an appropriate physical examination. Further routine diagnostic tests may also be performed to determine eligibility for approved studies. The tests and procedures are of minimal risk. When the screening has been completed, subjects will be informed of the options available at the time for participation in available, approved research protocols.

ELIGIBILITY:
INCLUSION CRITERIA:

All patients who may be eligible for other currently approved protocols.

Inclusion and exclusion criteria will vary according to the protocol(s) for which the patient is being screened.

Patients may be eligible if they have rare, unusual, interesting or unknown conditions that require diagnosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2000-01; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States